CLINICAL TRIAL: NCT03783455
Title: Assessment of Short-term Effectiveness of Five Local Treatment Modalities in Patients With Symptomatic Knee Osteoarthritis: a Randomized Prospective Study
Brief Title: Effectiveness of Five Intraarticular Strategies on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAJL
Record Dates: First submitted 2018-12-13; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Osteo Arthritis Knee
Keywords: Corticosteroid; Hyaluronic acid; Joint Lavage
MeSH Terms: interventions — Adrenal Cortex Hormones; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Open, controlled, randomized and prospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Non arthroscopic joint lavage (NAJL) (Active Comparator): Establishment of sterile areas and cleaning of the skin around the knee with a povidone-iodine solution, followed by an injection of local anesthetic (5 mL of 2% mepivacaine hydrochloride) into the outer mediopatellar zone. The anesthetic was allowed to act, and an access way was then opened with a No. 16 abocat. Any effusion in the joint was drained. Then, approximately 100 mL of cold saline was instilled through the outer access way. Once the knee was distended, a further 5 mL of local anesthetic was injected into the inner mediopatellar zone, and a new abocat guide was used to establish the inner drainage way. The lavage proper involved instillation of 4 L of cold (8ºC) saline at a constant flow-rate using a dropper line connected to the entry way; the inner zone was also connected to another, free-fall dropper.
  Interventions: Procedure: Non arthroscopic joint lavage
- Non arthroscopic joint lavage plus corticosteroid (Active Comparator): Establishment of sterile areas and cleaning of the skin around the knee with a povidone-iodine solution, followed by an injection of local anesthetic (5 mL of 2% mepivacaine hydrochloride) into the outer mediopatellar zone. The anesthetic was allowed to act, and an access way was then opened with a No. 16 abocat. Any effusion in the joint was drained. Then, approximately 100 mL of cold saline was instilled through the outer access way. Once the knee was distended, a further 5 mL of local anesthetic was injected into the inner mediopatellar zone, and a new abocat guide was used to establish the inner drainage way. The lavage proper involved instillation of 4 L of cold (8ºC) saline at a constant flow-rate using a dropper line connected to the entry way; the inner zone was also connected to another, free-fall dropper. Following administration of the joint lavage, the NAJL plus corticosteroid group was given an intra-articular injection containing 40 mg of triamcinolone acetonide.
  Interventions: Procedure: Non arthroscopic joint lavage plus corticosteroid
- Non arthroscopic joint lavage plus hyaluronic acid (Active Comparator): Establishment of sterile areas and cleaning of the skin around the knee with a povidone-iodine solution, followed by an injection of local anesthetic (5 mL of 2% mepivacaine hydrochloride) into the outer mediopatellar zone. The anesthetic was allowed to act, and an access way was then opened with a No. 16 abocat. Any effusion in the joint was drained. Then, approximately 100 mL of cold saline was instilled through the outer access way. Once the knee was distended, a further 5 mL of local anesthetic was injected into the inner mediopatellar zone, and a new abocat guide was used to establish the inner drainage way. The lavage proper involved instillation of 4 L of cold (8ºC) saline at a constant flow-rate using a dropper line connected to the entry way; the inner zone was also connected to another, free-fall dropper. Following administration of the joint lavage, the patients were given an intra-articular injection containing 4 ml of a bioengineered hyaluronic acid.
  Interventions: Procedure: Non arthroscopic joint lavage plus hyaluronic acid
- Intraarticular injection of hyaluronic acid (Active Comparator): Establishment of sterile areas and cleaning of the skin around the knee with a povidone-iodine solution. This was followed by an intraarticular injection containing 4 mL of a bioengineered hyaluronic acid.
  Interventions: Procedure: Intraarticular injection of hyaluronic acid
- Intraarticular injection of corticosteroid (Active Comparator): Establishment of sterile areas and cleaning of the skin around the knee with a povidone-iodine solution. This was followed by an intraarticular injection containing 40 mg of triamcinolone acetonide.
  Interventions: Procedure: Intraarticular injection of corticosteroid

INTERVENTIONS:
Procedure: Non arthroscopic joint lavage — Instillation of 4 litters of cold physiological serum
  Other Names: NAJL
  Arms: Non arthroscopic joint lavage (NAJL)
Procedure: Non arthroscopic joint lavage plus corticosteroid — Instillation of 4 litters of cold physiological serum followed by intraarticular injection of triamcinolone
  Arms: Non arthroscopic joint lavage plus corticosteroid
Procedure: Non arthroscopic joint lavage plus hyaluronic acid — Instillation of 4 litters of cold physiological serum followed by intraarticular injection of hyaluronic acid
  Arms: Non arthroscopic joint lavage plus hyaluronic acid
Procedure: Intraarticular injection of corticosteroid — Intraarticular injection containing 40 mg of triamcinolone acetonide.
  Arms: Intraarticular injection of corticosteroid
Procedure: Intraarticular injection of hyaluronic acid — Intraarticular injection containing 4 mL of a bioengineered hyaluronic acid.
  Arms: Intraarticular injection of hyaluronic acid

SUMMARY:
BACKGROUND: Current medical treatment strategies for knee osteoarthritis (OA) are aimed at pain reduction and symptom control. The Non-Arthroscopic Joint Lavage (NAJL) is included inside the therapeutic algorithm of knee OA when other therapies are contraindicated or have lost effectiveness. The large variety of potentially invasive interventions available (joint lavage included) has raised the need to assess their efficacy. The objective of this study is to compare the short-term effectiveness of five treatment strategies in patients with knee osteoarthritis (OA).

METHODS: It was conducted a randomized prospective study involving 150 patients of whom 76.7% were females. The age range was 40-81 years. All patients had knee OA according to the American College of Rheumatology criteria, with Kellgren-Lawrence radiographic grades II and III. Patients were assigned to five groups, 1) non-arthroscopic joint lavage (NAJL) (n= 30), 2) NAJL plus hyaluronic acid (HA) (n= 32), 3) NAJL plus corticosteroid (CS) (n= 32), 4) HA (n= 31), 5) CS (n= 25). Evaluations took place at baseline, one and three months after enrollment. Demographic variables, Western Ontario and McMaster University Osteoarthritis Index (WOMAC) and Lequesne scores were recorded. Statistical analysis included mixed analysis of variance, post-hoc comparisons with Sidak's adjustment, and multiple linear regression using as outcome WOMAC total at 3 months.

TRIAL REGISTRATION: The protocol of the study was approved by the "Hospital Universitario Reina Sofía" Ethics Committee, under the number 1996, in the Minutes 208 of 29 May 2012.

ELIGIBILITY:
Inclusion Criteria:

* Meeting American College of Rheumatology (ACR) criteria for knee OA, symptoms for at least three months despite conservative medical treatment, knee OA grade II or III on the radiological Kellgren-Lawrence scale, and voluntary collaboration.

Exclusion Criteria:

* ankylosis of joint;
* total arthroplasty or previous osteotomy
* infected injury;
* treatment with dicumarinic drugs or alterations in blood coagulation,
* venous insufficiency or episode of venous thrombosis;
* administration of hyaluronic acid (HA) in the previous year, and/or corticosteroid (CS) infiltration or NAJL in the previous three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
WOMAC 3.1 Index total | WOMAC total at 3 months
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.

SECONDARY OUTCOMES:
Lequesne Index | baseline, at one month and at three months
  Lequesne Index is a ten question questionnaire that asseses pain and function in patients with osteoarthritis of the knee. It is composed by five questions about pain, being three of them from 0 to 2, and two of them from 0 to 1 point, two questions about maximum distance walked (from 0 to 6 points one and from 0 to 2 the second) and four questions about activities of daily living (from 0 to 2). The total values is the sum of all questions points and range from 1 to 24, being 1-4 mild handicap, 5-7 moderate, 8-10 severe, 11-13 very severe, and >14 extremely severe handicap.
WOMAC 3.1 Index pain | WOMAC pain at baseline
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index pain | WOMAC pain at one month
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index pain | WOMAC pain at three months
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index function | WOMAC function at baseline
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index function | WOMAC function at one month
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index function | WOMAC function at three months
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index stiffness | WOMAC stiffness at baseline
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index stiffness | WOMAC stiffness at one month
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index stiffness | WOMAC stiffness at three months
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index total | WOMAC total at baseline
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
WOMAC 3.1 Index total | WOMAC total at one month
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. It can be used to monitor the course of the disease or to determine the effectiveness of anti-rheumatic medications. In the study it was used the validated Spanish version of the 5-point adjectival scale format (possible answers are none -0 points-, slight -1 point-, moderate -2 points-, severe -3 points- and extreme -4 points-). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Ladehesa, MD, Principal Investigator — Hospital Universitario Reina Sofía

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cope PJ, Ourradi K, Li Y, Sharif M. Models of osteoarthritis: the good, the bad and the promising. Osteoarthritis Cartilage. 2019 Feb;27(2):230-239. doi: 10.1016/j.joca.2018.09.016. Epub 2018 Oct 25. PMID 30391394
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Cooper C, Rannou F, Richette P, Bruyere O, Al-Daghri N, Altman RD, Brandi ML, Collaud Basset S, Herrero-Beaumont G, Migliore A, Pavelka K, Uebelhart D, Reginster JY. Use of Intraarticular Hyaluronic Acid in the Management of Knee Osteoarthritis in Clinical Practice. Arthritis Care Res (Hoboken). 2017 Sep;69(9):1287-1296. doi: 10.1002/acr.23204. Epub 2017 Aug 8. No abstract available. PMID 28118523
- [Background] Escobar A, Quintana JM, Bilbao A, Azkarate J, Guenaga JI. Validation of the Spanish version of the WOMAC questionnaire for patients with hip or knee osteoarthritis. Western Ontario and McMaster Universities Osteoarthritis Index. Clin Rheumatol. 2002 Nov;21(6):466-71. doi: 10.1007/s100670200117. PMID 12447629